CLINICAL TRIAL: NCT05423574
Title: Feasibility Study of Robotic Trans-Abdominal Retromuscular Umbilical Prosthesis (r-TARUP) for the Treatment of Primary and Incisional Ventral Hernia
Brief Title: Robotic Trans-Abdominal Retromuscular Umbilical Prosthesis (r-TARUP)
Acronym: r-TARUP
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI130
Record Dates: First submitted 2021-09-13; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-08

CONDITIONS: Ventral Hernia
Keywords: robotic assisted laparoscopy
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: robotic Trans Abdomino Pre Peritoneal prothesis repair — The treatment of primary and incisional ventral hernia using the robotic assisted laparoscopy technique

SUMMARY:
Combining the advantage of minimally invasive surgery with laparoscopy to reduce postoperative complications and the placement of a retromuscular prosthesis with closure of the defect in order to reduce the risk of adhesion and restore normal anatomy in the treatment of primary and incisional ventral hernias, is made possible through robotic assistance.

The challenge of this study concerns the evaluation of quality of life, postoperative pain and recurrence at 6 months in the management of primary and incisional ventral hernias by robot-assisted laparoscopic approach.

DETAILED DESCRIPTION:
The robotic-assisted laparoscopic approach for the treatment of primary and secondary ventral hernias is already used in the visceral department of Nancy in France. This technique seems to reduce post operative pain, to improve quality of live and to reduce recurrence. The goal of the study is to evaluate the benefices of this technique. The quality of life, postoperative pain and recurrence will be evaluated at one and six months postoperatively. The recurrence will be evaluated by clinical examination and a computed tomography scan performed at sixth month postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* major patients undergoing a robotic-assisted laparoscopy procedure for the treatment of ventral hernia repair

Exclusion Criteria:

* patient minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients undergoing a robotic-assisted laparoscopy procedure for the treatment of ventral hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 6 months | 6 months
  Evaluated by clinical examination

SECONDARY OUTCOMES:
Post operative pain | 6 months
  Evaluated by a digital scale, from 0 (no pain) to 10 (maximal pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire (CHRU), Nancy, France